CLINICAL TRIAL: NCT02226367
Title: Prazosin Augmentation of Outpatient Treatment of Alcohol Use Disorders in Active Duty Soldiers With and Without PTSD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seattle Institute for Biomedical and Clinical Research (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency); VA Puget Sound Health Care System (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: W81XWH-12-2-0094
Record Dates: First submitted 2014-07-15; First posted 2014-08-27 (Estimated); Results first posted 2023-02-03 (Actual); Last update posted 2023-02-03 (Actual); Status verified 2023-01

CONDITIONS: Alcohol Use Disorders; Stress Disorders, Posttraumatic; Combat Disorders
Keywords: prazosin; alcohol use disorders; posttraumatic stress disorder; PTSD; combat trauma; military; alpha-1 adrenoreceptor antagonist
MeSH Terms: conditions — Alcoholism; Stress Disorders, Post-Traumatic; Combat Disorders | interventions — Prazosin; Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- prazosin hydrochloride (Active Comparator): Prazosin hydrochloride taken orally. Titrated to a maximum dose 4 mg in the morning, 6 mg in the afternoon, and 10 mg at bedtime. (20 mg total daily at maximum dose) Dose increase will occur if the participant does not have unacceptable side effects.
  Interventions: Drug: prazosin hydrochloride
- placebo (Placebo Comparator): Placebo. Oral capsule with comparable appearance to active treatment. Titrated in same manner as active treatment.
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: prazosin hydrochloride — study drug arm prazosin
  Other Names: prazosin; Pfizer Minipress
  Arms: prazosin hydrochloride
Drug: placebo — study drug arm placebo
  Other Names: sugar pill
  Arms: placebo

SUMMARY:
The purpose of the study is to evaluate if the drug prazosin:

* will decrease alcohol use in active duty members of the military who served in Iraq and/or Afghanistan and
* determine if presence or absence of posttraumatic stress disorder affects treatment.

DETAILED DESCRIPTION:
The proposed study is a 19-week, titration to stable dose, randomized, two-group parallel-design, double-blind, placebo-controlled trial to evaluate the efficacy of prazosin for decreasing alcohol use in 200 active duty Service Members who served in the conflicts in Iraq and/or Afghanistan who are receiving standard outpatient treatment for alcohol use disorders at Joint Base Lewis-McChord. Treatment groups will be stratified by presence or absence of posttraumatic stress disorder (PTSD) and by assignment to the 6-week or 12-week Army Substance Abuse Program. The hypotheses are that: 1) prazosin is more effective than placebo for alcohol use disorders in these Service Members; and 2) that prazosin effect size will be greater in Service Members with PTSD than without PTSD.

ELIGIBILITY:
Inclusion Criteria

* Male and female active duty returnees from the conflicts in Iraq and/or Afghanistan over the age of 21 with a current Diagnostic and Statistical Manual of Mental Disorders IV diagnosis of Alcohol Abuse or Dependence or a current Diagnostic and Statistical Manual of Mental Disorders 5 diagnosis of Alcohol Use Disorder
* Participant in Army Substance Abuse Program (6 or 12 week program)
* Recent alcohol consumption: more than 14 (women) or 21 (men) drinks per week for at least 2 weeks in the past 60 day period OR at least 2 days of heavy drinking in the past 60 day period (4 or more drinks for women and 5 or more drinks for men)
* Good general medical health (see Exclusion Criteria below)
* Women of childbearing potential must agree to abstain from sexual relations that could result in pregnancy or use an effective method of birth control acceptable to both participant and the study clinician during the study. Men are not required to use contraception during the study.
* Concomitant use of naltrexone and/or antabuse must be stable for 2 weeks prior to Baseline
* Capacity to provide informed consent
* English fluency

Exclusion Criteria

* Current diagnosis of opioid, methamphetamine, cocaine, marijuana, or other illegal substance dependence or abuse.
* Signs or symptoms of alcohol withdrawal at the time of initial consent
* Current diagnosis of schizophrenia, other psychotic disorder, manic phase of bipolar disorder, or cognitive disorder.
* Suicide attempt or suicidal ideation with intent in the past month.
* Significant acute or chronic medical illness, including unstable angina, recent myocardial infarction, history of congestive heart failure, preexisting hypotension (systolic <100) or orthostatic hypotension (defined as a systolic drop > 20 mmHg after two minutes standing accompanied by lightheadedness or syncope); insulin-dependent diabetes mellitus; chronic renal or hepatic failure, acute pancreatitis, Meniere's disease. Liver function tests more than 5 times the upper limit.
* Concomitant use of trazodone (due to increased risk of priapism). There will be a two week trazodone washout period before the baseline visit.
* Concomitant use of an alpha-1 blocker medication or insulin
* Use of prazosin in the 4 weeks prior to Baseline.
* History of prazosin sensitivity/allergy

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 158 (Actual)
Dates: Start 2015-01; Primary Completion 2018-09-20 (Actual); Study Completion 2018-10-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Murray Raskind, MD, Principal Investigator — Department of Veterans Affairs Puget Sound Health Care System
Locations (1):
- Madigan Army Medical Center, Tacoma, Washington, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Active duty soldiers participating in command mandated Army outpatient alcohol treatment were randomized to the brain-penetrant alpha-1 adrenergic receptor antagonist prazosin or placebo for 13 weeks.
  The period of enrollment and completion of study procedures was January, 2015, through July, 2018.
  The study was ended following enrollment of 158 participants due to end of funding.
Period: Overall Study
Arm/Group | Prazosin Hydrochloride | Placebo
Started | 46 | 56
Completed | 37 | 49
Not Completed | 9 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Prazosin Hydrochloride | Placebo | Total
Number analyzed (Participants) | 46 | 56 | 102
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.2 (6.5) | 29.8 (6.8) | 29.6 (6.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 3 | 5
  Male | 44 | 53 | 97
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 8 | 15
  Not Hispanic or Latino | 38 | 47 | 85
  Unknown or Not Reported | 1 | 1 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 9 | 13
  White | 31 | 33 | 64
  More than one race | 4 | 6 | 10
  Unknown or Not Reported | 7 | 6 | 13
Region of Enrollment [Number; unit: participants]
  United States | 46 | 56 | 102

OUTCOME MEASURES:

1. Primary Outcome: Change in Penn Alcohol Craving Scale Score
Description: Penn Alcohol Craving Scale (PACS)
  The PACS is a self-report paper-and-pencil instrument. This five-item, self-report measure includes questions about the frequency, intensity, and duration of craving, the ability to resist drinking, and asks for an overall rating of craving for alcohol for the previous week. Each question is scaled from 0 to 6. Total scores are 0 to 30. Lower scores indicate less alcohol craving. Higher scores indicate more alcohol craving.
Time Frame: Change at Week 13 from Baseline
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Prazosin Hydrochloride | Placebo
Number analyzed (Participants) | 46 | 56
units on a scale | 7.4 (4.1) | 8.8 (6.4)

ADVERSE EVENTS:
Time Frame: Adverse events were tracked from initiation of study drug until 30 days following study completion or termination. approximately 23 weeks.
Description: This study utilized an Adverse Events Checklist of anticipated adverse events of prazosin, and open-ended adverse event reporting.
Arm/Group | Prazosin Hydrochloride | Placebo
All-Cause Mortality (participants affected / at risk) | 0/46 | 0/56
Serious Adverse Events (participants affected / at risk) | 2/46 | 1/56
Other Adverse Events (participants affected / at risk) | 44/46 | 52/56
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Prazosin Hydrochloride (N=46) | Placebo (N=56)
skull fracture and subdural hematoma (General disorders) | 0 | 1 — One participant randomized to placebo suffered a fractured skull and subdural hematoma resulting from a fall while alcohol intoxicated.
Suicidal Ideation (Psychiatric disorders) | 1 | 0 — One participant was psychiatrically hospitalized for suicidal ideation.
anxiety associated with occupational stressors (Psychiatric disorders) | 1 | 0 — One participant was hospitalized due to anxiety associated with occupational stressors.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Prazosin Hydrochloride (N=46) | Placebo (N=56)
dizziness on standing (General disorders) | 18 | 9
Nasal Congestion (General disorders) | 24 | 18
Nausea (Gastrointestinal disorders) | 14 | 8
Lightheadedness (General disorders) | 22 | 16
Weakness (General disorders) | 10 | 6
Palpitations (Cardiac disorders) | 8 | 5
Peripheral edema (General disorders) | 1 | 4
Depressed Mood (Psychiatric disorders) | 3 | 14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-02-26): https://cdn.clinicaltrials.gov/large-docs/67/NCT02226367/Prot_SAP_000.pdf